CLINICAL TRIAL: NCT04859075
Title: Efficacy and Safety of Alflorex® Bei Reizdarm, a Probiotic Containing Bifidobacterium Longum 35624®, in Patients With Irritable Bowel Syndrome in Medical Practice
Brief Title: Efficacy and Safety of Alflorex Bei Reizdarm in Patients With Irritable Bowel Syndrome
Status: Terminated | Type: Observational
Why Stopped: economic reasons
Sponsor: Medice Arzneimittel Pütter GmbH & Co KG (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: 6630-0280-01
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Bifidobacterium longum 35624 — 1 capsule daily

SUMMARY:
This Post-Market Clinical-Follow Up (PMCF) study gains data on the efficacy and safety of "Alflorex bei Reizdarm", a probiotic based on Bifidobacterium longum 35624, in the daily use by irritable bowel syndrome (IBS) patients. The aim of this study is the observation of the influence of "Alflorex bei Reizdarm" on typical symptoms, severity score and quality of life of IBS patients in medical practice and everyday use.

DETAILED DESCRIPTION:
This Post-Market Clinical-Follow Up (PMCF) study observes adult patients with irritable bowel syndrome (IBS) which receive "Alflorex bei Reizdarm", a probiotic based on Bifidobacterium longum 35624, for 8 weeks by recommendation of their physician. IBS symptoms are recorded on a weekly basis by the participants. IBS severity score, interference with general life and safety parameters are also recorded. Primary objective is the assessment of the change in overall IBS symptoms (sum of abdominal pain, bloating, gas, difficulty in defecating/constipation and urgency/diarrhoea).

ELIGIBILITY:
Inclusion Criteria:

Adult, diagnosed IBS patients with typical IBS symptoms (abdominal pain, bloating, gas, constipation or diarrhea) and physician's recommendation to take the study medication (probiotic with B. longum 35624) for 8 weeks

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBS patients of general practicioners and gastroenterologists
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Relative change in overall IBS symptoms compared to day 1 (sum of abdominal pain, bloating, gas, difficulty in defecating/constipation and urgency/diarrhoea symptom scores) | assessed weekly over 8 weeks (from day 1 to day 57)
  rated by participant on a 6-point Likert scale (from 0 "no symptoms" to 5 "very severe")

SECONDARY OUTCOMES:
Relative change in the individual IBS symptoms abdominal pain, gas, bloating, difficulty in defecating/constipation and urgency/diarrhoea compared to day 1 | assessed weekly over 8 weeks (from day 1 to day 57)
  rated by participant on a 6-point Likert scale (from 0 "no symptoms" to 5 "very severe")
Severity score of irritable bowel syndrome compared to day 1 | assessed at day 1, day 29 and day 57
  German IBS severity scoring system questionnaire by the participant (IBS-SSS, scoring from 0 to 500; higher scores indicating higher severity of IBS symptoms)
Efficacy & tolerability by physician | assessed at day 57
  rated on a 6-point Likert scale (from 1 "very good" to 6 "unsatisfactory")
Efficacy & tolerability by participant | assessed at day 57
  rated on a 6-point Likert scale (from 1 "very good" to 6 "unsatisfactory")
Interference of IBS symptoms with general life | assessed at day 1, day 29 and day 57
  rated by the participant by question 5 of the German IBS-SSS questionnaire (scoring from 0 to 100; higher scores indicating higher interference with general life)

CONTACTS AND LOCATIONS:
Locations (1):
- Several General Practicioner and Gastroenterologists (Multicentric), Düsseldorf, North Rhine-Westphalia, Germany